CLINICAL TRIAL: NCT04694066
Title: Qigong for Pre-frail and Frail Older Cancer Survivors: A Pilot Randomized Controlled Trial
Brief Title: Qigong for Pre-frail and Frail Older Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Cheung Shuk-Ting, Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HKUCTR-2708
Record Dates: First submitted 2020-12-30; First posted 2021-01-05 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Cancer; Frailty
Keywords: Frailty; Cancer survivors; Qigong; Feasibility
MeSH Terms: conditions — Neoplasms; Frailty | interventions — Qigong

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The care providers, though cannot be blinded, will not have knowledge about the aims of the study. The research assistants responsible for assessing the outcomes and entering the data will be blinded to the group.
  allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Qigong (Experimental): The entire intervention will last 16 weeks, including 1-hour supervised training sessions twice a week during weeks 1 to 8 (training; 16 hours), and 1-hour supervised weekly follow-up sessions during weeks 9 to 16 (followup; 8 hours). The sessions will be supervised by an experienced qigong master.
  Interventions: Behavioral: Qigong
- Light flexibility exercise (Active Comparator): The control group will practice light flexibility exercise only, with the same duration and frequency of supervised sessions identical to the qigong sessions. The supervised sessions will be conducted by a certified exercise trainer.
  Interventions: Behavioral: Light flexibility exercise

INTERVENTIONS:
Behavioral: Qigong — Qigong Baduanjin, comprising eight standardized movements, will be adopted in the study. It is practiced as a combination of body movements, breath control, and mindful meditation.
  Arms: Qigong
Behavioral: Light flexibility exercise — The supervised sessions will include seated and standing stretches that target upper (neck, arms, upper back, shoulders, and chest) and lower body (quadriceps, hamstrings, calves, and hips), as well as trunk rotations.
  Arms: Light flexibility exercise

SUMMARY:
To-date, there is no evidence on qigong's effects for improving well-being of pre-frail and frail older cancer survivors. Our aim is to conduct a pilot study for testing out the feasibility and acceptability of a qigong intervention to the elderly cancer survivors.

DETAILED DESCRIPTION:
Frailty is an emerging concept in geriatric research and practice. It is defined as a state of increased vulnerability to adverse outcomes including death. A cohort study has found that respondents with cancer were significantly more frail compared to those without cancer. A plausible explanation is both cancer itself and the therapies used to treat it add additional stressors that challenge a patient's physiologic reserve. A systematic review has revealed a high prevalence of frailty and pre-frailty in older cancer patients, with the median estimates of 42% and 43%, respectively. Cancer treatment can hasten survivors' aging process and increase their risk of developing frailty, thus placing cancer survivors at heightened risk of such poor health outcomes as falls, fractures, and disability. This calls for effective interventions that would improve frailty in older cancer survivors.

Qigong, a type of mind-body intervention, is particularly suitable for older adults, as it is implemented without aerobic and musculoskeletal strain. This equipment-free form of exercise is ideal for settings with limited resources, as well as for the frail elderly, because it can be performed at home at any time, reducing such barriers as weather, transportation, and cost. Meta-analysis suggests that Baduanjin is beneficial in the general population in terms of improved quality of life, balance, handgrip strength, and trunk flexibility. To our knowledge, there is no evidence on qigong's effects for improving well-being of pre-frail and frail older cancer survivors. Our aim is therefore to conduct a pilot study for testing out the feasibility and acceptability of a qigong intervention to the elderly cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

1. aged ≥65
2. diagnosed with stage I-III non-metastatic cancer
3. completed primary treatment with curative intent (surgery, chemotherapy, and/or radiation therapy) 6 months to 5 years prior to baseline assessments with no recurrence or occurrence of additional cancers
4. classified as pre-frail or frail based on Fried frailty criteria
5. can communicate in Cantonese or Putonghua
6. written informed consent

Exclusion Criteria:

1. regular qigong training or other mind body intervention (once or more per week) within the previous 6 months
2. medical conditions affecting mobility, predisposing to falls, or precluding qigong practice (e.g., neurological disease, musculoskeletal disorder, recent myocardial infarction, breathing difficulties requiring oxygen)

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Feasibility: Study completion rate | 16 weeks
  The proportion of participants who completed the data collection among those randomized will be recorded at each time point.
Feasibility: Attendance rate | 16 weeks
  Participants' attendance to the supervised sessions will be recorded at each time point.

SECONDARY OUTCOMES:
Change in frailty status | study entry, 8 weeks, 16 weeks
  Participants' frailty status will be assessed using the Fried frailty criteria, which consists of 5 criteria: slowness , weakness , unintentional weight loss , exhaustion and low activity.
Change in Short Physical Performance Battery scores | study entry, 8 weeks, 16 weeks
  Short Physical Performance Battery is an objective assessment tool used to measure the physical performance of participants in three functional tasks.
Change in Short-Form Geriatric Depression Scale scores | study entry, 8 weeks, 16 weeks
  The Short-Form Geriatric Depression Scale (15 items) will be used to measure psychological well-being. Scores range from 0 to 15, with higher scores representing more severe depressive symptoms.
Change in European Organization for Research and Treatment of Cancer Quality of Life Core Questionnaire-C30 scores | study entry, 8 weeks, 16 weeks
  European Organization for Research and Treatment of Cancer Quality of Life Core Questionnaire-C30 (30 items) will be used to assess health-related quality of life specifically in cancer patients. The questionnaire is composed of five functional scales, three symptom scales, a global health status / QoL scale, and six single items. scale. Scores of all subscales and single-item measures range from 0 to 100. Higher scores for functional scales represent higher level of functioning, global health status/quality of life, but higher scores for a symptom scale / item represent a higher level of symptom severity.
Change in Modified Barthel Index scores | study entry, 8 weeks, 16 weeks
  The Modified Barthel Index will be used to measure participants' performance in activities of daily living such as eating, personal hygiene, and bathing, rated on an arbitrary 2- to 4-point scale depending on the amount of assistance needed. Scores range from 0 (an inability to perform) to 15 (total independence).

CONTACTS AND LOCATIONS:
Overall Officials: Denise Cheung, Principal Investigator — The University of Hong Kong
Locations (2):
- Hong Kong (2):
  - Queen Mary Hospital, Hong Kong
  - Pamela Youde Nethersole Eastern Hospital, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
Data may be available upon reasonable request.

REFERENCES:
- [Derived] Cheung DST, Chau PH, Lam TC, Ng AYM, Kwok TWH, Takemura N, Woo J, Yu DS, Lin CC. A pilot randomized controlled trial using Baduanjin qigong to reverse frailty status among post-treatment older cancer survivors. J Geriatr Oncol. 2022 Jun;13(5):682-690. doi: 10.1016/j.jgo.2022.02.014. Epub 2022 Mar 7. PMID 35272982